CLINICAL TRIAL: NCT03737292
Title: Comparison of Plasma Concentration And Efficacy Of Liposomal Bupivacaine And Plain Bupivacaine After Intercostal Injections For Pain Management After Thoracoscopy
Brief Title: Liposomal Bupivacaine Versus Plain Bupivacaine After Intercostal Injections For Pain Management After Thoracoscopy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Zoulfira Nisnevitch-Savarese, Assistant Professor of Anesthesiology & Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10129
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Pharmacokinetics
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled, double blind study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exparel (Experimental): Intercostal injection of 266mg of Exparel diluted to 30 ml.
  Interventions: Drug: Exparel
- Bupivacaine (Active Comparator): Intercostal injection of 0.5% Bupivacaine 2 mg/kg dose diluted to 30 ml.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel — The intercostal blocks will be performed at several levels corresponding to the incisions and chest tube insertion sites + two levels above and two levels below the incisions. On average, 5-6 intercostal spaces will be injected with 4-5 ml of local anesthetic at each level.
  Arms: Exparel
Drug: Bupivacaine — The intercostal injections of 0.5% Bupivacaine 2 mg/kg dose diluted to 30 ml total will be performed at several levels corresponding to the incisions and chest tube insertion sites + two levels above and two levels below the incisions.
  Arms: Bupivacaine

SUMMARY:
The purpose of this study is to assess pharmacokinetics of liposomal bupivacaine (Exparel) after multilevel intercostal injections of this local anesthetic for pain control during and after thoracoscopic surgeries.

The specific aim of this study is to evaluate plasma concentration of bupivacaine after intraoperative intercostal injections of 266 mg of liposomal bupivacaine and compare it to plasma concentrations of bupivacaine after intercostal injections of 2mg/kg of 0.5% plain Bupivacaine with maximal dose of 30 ml or 150 mg.

The hypothesis of the study is that plasma concentration of bupivacaine after intercostal injections of 266 mg of liposomal bupivacaine will be similar to concentrations after injections of plain bupivacaine, and will remain below the toxic level threshold range of 2000-3000 ng/mL (2-3 mg/L) at which central nervous system and cardiovascular adverse events would be expected to occur.

The secondary objective is to evaluate if intercostal injections of 266 mg of liposomal bupivacaine will significantly reduce opioid consumption and postsurgical pain, within the first 48 hours and up to 3 months after minimally invasive thoracic surgeries, to determine if both acute and chronic post-thoracotomy pain can be decreased by intraoperative intercostal injections of liposomal bupivacaine.

Additionally, the rate of pneumonia, the rate of atrial fibrillation and length of hospital stay will be assessed as secondary outcomes after thoracic surgeries. These outcomes can be affected by the level of postoperative pain and inflammation.

Significance of this study: If positive, the results of this research have the potential to significantly improve pain management after thoracoscopic surgery.

Based on prior experience, prolonged analgesia after liposomal bupivacaine injection is safe, and may help reduce perioperative opioid consumption and decrease opioid related complications. It will improve patient comfort, eliminate need for indwelling neuraxial catheters and risks associated with them.

DETAILED DESCRIPTION:
Liposomal bupivacaine is a relatively new drug formulation. Its safety and side effect profile after intercostal injection has not been extensively studied. Most of the data comes from studies where the medicine was used for wound infiltrations and peripheral nerve blocks for orthopedic surgeries, or from preclinical volunteer studies. PK profile of Exparel varies significantly with different blocks and administration techniques. Very few data are available about pharmacokinetics of the drug after intercostal injections.

Because Exparel contains plain bupivacaine in a liposomal form, it allows for a slower release of the medication from the injection site into the blood stream, and prolongs the duration of action of this local anesthetic. During intercostal infiltration, a local anesthetic is injected into a highly vascular area with increased rate of intravascular absorption and potential risk of toxicity.

Also, because liposomal formulation provides a slow release of local anesthetic, the maximum recommended dose of Exparel (266mg) for intercostal injections is higher than a maximum recommended dose for plain bupivacaine (150mg), which can theoretically increase the risk of local anesthetic toxicity.

The plan of this s to analyze a pharmacokinetic profile and safety of liposomal bupivacaine compared with plain bupivacaine HCl. it is understood that absolute numbers can differ because the doses of the two formulations are different. Unfortunately, the dose of plain bupivacaine cannot be increased to match the dose of Exparel because of the risk of toxicity. The dose of Exparel should not be lowered, because lower doses have been shown to be less effective and are not clinically used at Hershey Medical Center.

Based on prior experience, it is known that prolonged analgesia after Exparel injection is safe, and can help reduce perioperative opioid consumption and decrease opioid related complications.

The goal of this study is to demonstrate that despite the higher total dose of bupivacaine administered via Exparel formulation as an intercostal injection, maximal plasma concentration will remain within therapeutic levels of 700-1,000 ng/mL, and below toxic level threshold range of 2000-3000 ng/mL at which central nervous system and cardiovascular adverse events would be expected to occur. As a result, many more patients in the future can benefit from a wider use of Exparel for pain management after thoracic surgeries.

Pneumonia and atrial fibrillation are well known complications of thoracic surgeries. The etiology of atrial fibrillation after lung resection involves a combination of postoperative hyperadrenergic activity and atrial dilatation. Increased vagal tone, atrial inflammation, pulmonary hypertension, hypoxemia, or infection may also contribute. Preclinical studies have shown a multitude of interactions between local anesthetics and the inflammatory system. It is known that proinflammatory effects are attenuated by perioperative intravenous lidocaine infusion via blocking the process of priming of polymorphonuclear granulocytes (PMN). Since pneumonia and atrial fibrillation after thoracic surgery can be attributed in part to inflammation, the hypothesis is that liposomal bupivacaine, due to higher concentration and longer duration of action, can decrease incidence of these complications and improve hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over age 18 undergoing minimally invasive thoracic surgeries including but not limited to:

1. VATS wedge resection /segmentectomy
2. VATS lobectomy.
3. Robot assisted thoracoscopic wedge resection/segmentectomy.
4. Robot assisted thoracoscopic lobectomy procedures.

Exclusion Criteria:

1. Patients under18 years of age
2. Patients weighing less than 48 kg
3. Pregnant and lactating females will be excluded from the trial
4. Patients preoperatively taking narcotics for chronic pain in proximity to surgical site
5. Patients with previous ipsilateral thoracic surgery
6. Patients undergoing pleurectomy/mechanical pleurodesis.
7. Patients with high likelihood of conversion from thoracoscopic procedure to open thoracotomy as determined by an operating surgeon
8. Patients with pre-existing painful conditions (CRIPS, fibromyalgia, neuropathy)
9. Patients unable to reliably communicate pain scores such as patients with dementia, alterations in mental status
10. Patients with hypersensitivity to local anesthetics and pain medications used in the study
11. Patients with previous thoracic spine surgeries
12. Patients with increased creatinine (over 1.5mg/dl)
13. Patients with liver dysfunction
14. Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of bupivacaine | 0.5, 1, 2, 4, 8, 12, 24, 32, 48, 72 hours after intraoperative multiple level intercostal injections.
  The primary end points to be measured in the study are plasma concentrations of bupivacaine 0.5, 1, 2, 4, 8, 12, 24, 32, 48 hours after intraoperative multiple level intercostal injections of plain Bupivacaine or Exparel. If the patient remains in the hospital, additional samples will be collected at 72 hours. If the patient gets discharged before this time, the last sample will be drawn at time of discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Zoulfira Nisnevitch-Savarese, MD, Principal Investigator — Penn State Hershey College of Medicine
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott DB. Evaluation of the toxicity of local anaesthetic agents in man. Br J Anaesth. 1975 Jan;47(1):56-61. doi: 10.1093/bja/47.1.56. PMID 1096908
- [Background] Richard BM, Rickert DE, Doolittle D, Mize A, Liu J, Lawson CF. Pharmacokinetic Compatibility Study of Lidocaine with EXPAREL in Yucatan Miniature Pigs. ISRN Pharm. 2011;2011:582351. doi: 10.5402/2011/582351. Epub 2011 Dec 27. PMID 22389853
- [Background] Scott DB, Lee A, Fagan D, Bowler GM, Bloomfield P, Lundh R. Acute toxicity of ropivacaine compared with that of bupivacaine. Anesth Analg. 1989 Nov;69(5):563-9. PMID 2679230
- [Background] Knudsen K, Beckman Suurkula M, Blomberg S, Sjovall J, Edvardsson N. Central nervous and cardiovascular effects of i.v. infusions of ropivacaine, bupivacaine and placebo in volunteers. Br J Anaesth. 1997 May;78(5):507-14. doi: 10.1093/bja/78.5.507. PMID 9175963
- [Background] Neal JM, Barrington MJ, Fettiplace MR, Gitman M, Memtsoudis SG, Morwald EE, Rubin DS, Weinberg G. The Third American Society of Regional Anesthesia and Pain Medicine Practice Advisory on Local Anesthetic Systemic Toxicity: Executive Summary 2017. Reg Anesth Pain Med. 2018 Feb;43(2):113-123. doi: 10.1097/AAP.0000000000000720. PMID 29356773
- [Background] Khalil KG, Boutrous ML, Irani AD, Miller CC 3rd, Pawelek TR, Estrera AL, Safi HJ. Operative Intercostal Nerve Blocks With Long-Acting Bupivacaine Liposome for Pain Control After Thoracotomy. Ann Thorac Surg. 2015 Dec;100(6):2013-8. doi: 10.1016/j.athoracsur.2015.08.017. Epub 2015 Oct 24. PMID 26507422
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739